CLINICAL TRIAL: NCT02819180
Title: Prospective Cohort Study to Evaluate Safety and Immunogenicity of Butantan Seasonal
Brief Title: Study to Evaluate Safety and Immunogenicity of Butantan Seasonal Influenza Vaccine - FLU-02-IB
Acronym: FLU-02-IB
Status: Completed | Type: Observational
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: FLU-02-IB
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines, Inactivated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy adults group: Healthy men and women between 18 and 59 years of age.
  Interventions: Biological: Butantan Influenza Trivalent, Fragmented and Inactivated vaccine
- Elderly group: Elderly over 60 years old.
  Interventions: Biological: Butantan Influenza Trivalent, Fragmented and Inactivated vaccine

INTERVENTIONS:
Biological: Butantan Influenza Trivalent, Fragmented and Inactivated vaccine
  Other Names: Butantan Influenza vaccine

SUMMARY:
Prospective cohort study to evaluate the safety and immunogenicity of the Butantan Influenza vaccine (Fragmented and Inactivated) among healthy adults with 18 to 59 years of age and elderly older than 60 years of age.

DETAILED DESCRIPTION:
Prospective cohort study to assess safety of one dose of theButantan Influenza vaccine (Fragmented and Inactivated) in the first 3 days after vaccination and its immunogenicity 21 days after vaccination among healthy adults with 18 to 59 years of age and elderly older than 60 years of age..

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, male or female aged 18 to 59
* Elderly aged 60 years completed and above
* To be available to participate in the study throughout its duration (approximately 21 days)
* To have medical indication to be vaccinated against influenza
* To demonstrate intention to participate in the study, as documented by signature in the study´s informed consent form.

Exclusion Criteria:

* Evidence of active neurological, cardiac, pulmonary, hepatic or renal disease as clinical history and/or physical examination (except hypertension under control among the elderly)
* Compromised immune system diseases including: HIV, diabetes mellitus, cancer (except basal cell carcinoma) and autoimmune diseases
* Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements
* Abusive usage of alcohol or drugs in the past 12 months that has caused medical, professional or family problems, indicated by clinical history
* Known systemic hypersensitivity to eggs or to any component of the vaccine
* History of severe adverse reaction after previous administration of an Influenza vaccine within 6 weeks following vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health adults with age between 18 and 59 years, as well as elderly over 60 years of age may participate in the study. To be included in the study, participants need to meet all inclusion criteria, and not fulfill any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Adverse events in the first 3 days post vaccination (Safety) | Three days
  Solicited and unsolicited local and systemic adverse reactions reported by the participants until Day 3 after vaccination.
Antibody response to each of the vaccine strains 21 days post vaccination (Immunogenicity) | 21 days
  Antibody response to each of the vaccine´s strains as measured by:
  * % seroconversion and/or
  * increase in the geometric mean of hemagglutination inhibition (HAI) titers and/or
  * % seroprotection.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Referência de Imunobiológicos Especiais (CRIE) Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Mondini G, Braga PE, Lopes MH, Sartori AMC, Miyaji KT, Infante V, Randi BA, Timenetsky MDCST, Ferreira JCOA, Sakita NK, Precioso AR. Prospective cohort studies to evaluate the safety and immunogenicity of the 2013, 2014, and 2015 seasonal influenza vaccines produced by Instituto Butantan. Rev Inst Med Trop Sao Paulo. 2018 Jul 30;60:e37. doi: 10.1590/S1678-9946201860037. PMID 30066805